CLINICAL TRIAL: NCT04206501
Title: OptiVol for Precision Medical Management of Heart Failure
Acronym: (OPTIMED-HF)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to COVID Pandemic
Sponsor: University of Rochester (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Spencer Rosero, MD, Professor Medicine M&D-Cardiology Div, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00003638
Record Dates: First submitted 2019-12-10; First posted 2019-12-20 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Ischemic and Non-ischemic Cardiomyopathy
Keywords: ICD; OptiVol-Monitor; Cardiac Compass; Garmin Vivo Smart; Guideline Directed Medical Therapy
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ICM guided Medical Management Group (Experimental): A pre-specified management regimen based on standard clinical practice will be provided to the study team in which medical management including medication dosing (focusing on beta-blockers and diuretics) will be monitored and modified using Cardiac Implantable Electronic Devices (CIED) and OptiVol Monitor data. Based on CIED and patient engagement data, the study team will adjust medications and dosages, and optimize activity/exercise steps.
  Interventions: Device: Medtronic ICD with Opti Vol-Monitor
- Conventional Management Control Group (No Intervention): Non-study physicians will receive CIED/OptiVol data (as in usual care) and its use and the management strategy will be left to his/her discretion. To control for patient contact, patients in the conventional management group will have the same study visits as the interventional group and will include in-person device interrogation, and documentation of any medications changes.

INTERVENTIONS:
Device: Medtronic ICD with Opti Vol-Monitor — Physiologic and functional data from Cardiac Implantable Electronic Devices (CIEDs), including information on heart rate, activity, and fluid status derived from the OptiVol monitor, together with a concurrent patient engagement strategy through remote interactions, can be used to optimize the medical management of HF patients implanted with an ICD.
  Arms: ICM guided Medical Management Group

SUMMARY:
This clinical study is designed to show that a multidisciplinary team following a pre-specified standard of care medication decision model based on data from an implanted cardioverter device will increase the rate of change in Guideline Directed Medical Therapy (GDMT) in the intervention group compared to the conventional group in patients with ischemic and non-ischemic cardiomyopathies.

DETAILED DESCRIPTION:
Subjects in this study will be randomized (2:1) to an intervention group whose medical care will be guided by data from a cardiac implantable electronic device (CIED) including information on heart rate, activity, and fluid status derived from the OptiVol monitor versus a conventional management control group. Subjects will followed for 12 months with follow up contact for 6 consecutive months and a chart review at 12 months. The study population will include patients with ischemic and non-ischemic cardiomyopathy who have had an ICD implanted per standard of care guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age on the date of randomization
* ICD implantation per guidelines for primary prevention in patients with ischemic and non-ischemic cardiomyopathy ≥3 calendar months ago.
* SMART Phone or tablet with Bluetooth capability with internet access.
* No other identifiable reversible cause explaining the left ventricular dysfunction

Exclusion Criteria:

* CRT implanted
* LVEF>45% in the last echocardiogram or other clinic imaging study performed.
* Medtronic device generator and/or device components not implanted
* Unstable clinical condition, life threatening arrhythmia
* Heart failure hospitalization within the preceding 3 calendar months
* Cognitive impairment
* Severe renal dysfunction (eGFR < 30 ml/min/m2)
* Serious known concomitant disease with a lift expectancy of < 12 calendar months
* Non-ambulatory NYHA class IV
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spencer Z Rosero, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Roth GA, Poole JE, Zaha R, Zhou W, Skinner J, Morden NE. Use of Guideline-Directed Medications for Heart Failure Before Cardioverter-Defibrillator Implantation. J Am Coll Cardiol. 2016 Mar 8;67(9):1062-1069. doi: 10.1016/j.jacc.2015.12.046. PMID 26940927
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 patients were enrolled and randomized to either Conventional Medical Therapy vs. Intervention group
Period: Overall Study
Arm/Group | ICM Guided Medical Management Group | Conventional Management Control Group
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total participants analyzed is 7.
Groups:
- Total: Total of all reporting groups
Arm/Group | ICM Guided Medical Management Group | Conventional Management Control Group | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13.6) | 65.7 (4.1) | 64 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7
History of Atrial Fibrillation [Count of Participants; unit: Participants] | 3 | 2 | 5
Ventricular Arrhythmias [Count of Participants; unit: Participants] | 3 | 1 | 4
NYHA Class 2 [Count of Participants; unit: Participants] — Number of participants with New York Heart Association Class 2. The NYHA classification ranges from a minimum of 1 to a maximum of 4. A higher score is associated with worsened outcomes.
  Participants | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Change in Medical Management With Beta-blockers, Diuretics and Sacubitril/Valsartan (Defined as Initiation, Termination, Switch, or Dosing Adjustment) in the Intervention Group Compared to Usual Care
Description: The rate of change as measured in the number of medications modified during medical management with beta-blockers, diuretics and sacubitril/Valsartan (defined as initiation, termination, switch, or dosing adjustment) in the intervention group compared to usual care will serve as the primary outcome. The (minimum, maximum) values (0,5) and the range (0 - 5) apply to the rate of change of the prespecified medications. The greater the rate of change, the more optimization (better) the intervention is altering medical management to personalize the regimen.
Time Frame: 6 Months
Population: The present study enrolled 7 patients randomized to ICM guided Medical Management Group or Conventional Management Control group
Measure: Mean (Standard Deviation); unit: Medications
Arm/Group | ICM Guided Medical Management Group | Conventional Management Control Group
Number analyzed (Participants) | 4 | 3
Medications | 3.3 (1.0) | 1.3 (1.2)
Statistical Analysis 1: Comparison: ICM Guided Medical Management Group vs Conventional Management Control Group; Due to the unexpected low enrollment during COVID pandemic, we aimed to primarily focus the limited analysis/description on the primary endpoint and exploratory analysis related to QOL; Test type: Superiority; p = 0.064, Chi-squared — The rate of change in HF medications (beta-blocker, diuretic, and Sacubitril/Valsartan) was compared betweenICM Guidedand usual care control group using chi-square analysis

2. Secondary Outcome: Mean Change in Quality of Life Score
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) was used to measure Quality of Life from index discharge to 6 months after discharge in the GDMT intervention vs. control (CMT) groups. Mean changes in KCCQ score for the overall summary score in which positive changes are associated with better QOL outcome and negative change associated with worsened outcome. The absolute KCCQ score can range from 0-100 with higher score associated with better outcomes.
Time Frame: 6 month
Population: Mean change in KCCQ overall summary score for each group. A positive change is associated with better outcome and a negative change in score is associated with worsening outcome on the KCCQ instrument. The range is 0-100 with a minimum of 0 and a maximum of 100.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ICM Guided Medical Management Group | Conventional Management Control Group
Number analyzed (Participants) | 4 | 3
score on a scale | 7.0 (15.8) | -9.4 (10.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ICM Guided Medical Management Group | Conventional Management Control Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICM Guided Medical Management Group (N=4) | Conventional Management Control Group (N=3)
Any Cardiac Related Event (Cardiac disorders) | 3 (7) | 2 (5) — Adverse Events were monitored/assessed as any cardiac related event without further specification.

LIMITATIONS AND CAVEATS:
Early termination due to COVID Pandemic leading to small numbers of subjects analyzed which limits interpretation of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT04206501/Prot_SAP_000.pdf